CLINICAL TRIAL: NCT04696068
Title: Impact on the Nutritional Status of Serving the Main Course on Porcelain Plates as a Replacement for Plastic Trays in Patients Over 65 Years of Age
Brief Title: Nutritional Status in Patients Over 65 Years of Age and Meal Presentation
Acronym: NUPOBA
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University Hospital, Caen (Other)
Responsible Party: Sponsor
Other Study IDs: 2020-A02315-34
Record Dates: First submitted 2021-01-04; First posted 2021-01-06 (Actual); Last update posted 2022-08-24 (Actual); Status verified 2022-07

CONDITIONS: ELDRELY
Keywords: malnutrition; aged; meal presentation; SEFI®; prealbumin
MeSH Terms: conditions — Malnutrition

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Control: The patients included in this group will receive meals with the usual presentation (plastic trays) during six days. Their data will be collected at day 1 and day 6.
- Experimental: The patients included in this group will receive the main course in porcelain plates during six days. Their data will be collected at day 1 and day 6.
  Interventions: Other: Porcelain plates

INTERVENTIONS:
Other: Porcelain plates — The patients will receive the same food in another presentation : porcelain plates instead of plastic trays
  Groups: Experimental

SUMMARY:
The prevalence of undernutrition in hospitals is estimated between 30 and 40% and up to 50% in the elderly. The consequences of undernutrition are significant: complications, delayed healing, higher risk of infections, pressure ulcers, lengthening of the length of stay, higher readmission rate, increased mortality, reduced quality of life, etc. In addition, the cost of hospital malnutrition is high for the health system. As a result, undernutrition is one of the axes of action of the french National Health Nutrition Program 2019-2023 (PNNS4). It can appear during hospitalization or be pre-existing and worsen during hospitalization. It is due to an unfavorable balance between expenditure and energy intake. One of the causes is incomplete consumption of meals served in hospital. Studies have shown that the appearance of the meal is a hindrance to patients feeding.

At the Caen Normandie University Hospital, meals have been served to patients in plastic trays for thirteen years. The presentation of the meals is a significant factor in not consuming meals in the hospital. In addition to the problem of the presentation of meals, plastic trays pose ergonomic problems: their height hinders the cutting and the gripping of food, which is difficult for patients with gripping problems; they can also be difficult to open for these same patients. They also pose environmental problems: the waste generated is not currently recycled.

The investigators hypothesize that presenting the main course on porcelain plates would reduce undernutrition and limit food waste.

The investigators therefore propose a study with the aim of:

* Compare the assessment of the perception of dietary intakes of patients receiving dishes presented on porcelain plates (experimental group) with that of patients receiving dishes in plastic trays (current system - control group) on D6 ± 1 day;
* Compare the evolution of indicators of nutritional status or risk in elderly patients receiving meals presented in porcelain plates (experimental group) compared to those receiving meals presented in plastic trays (control group);
* Evaluate food intake and food waste in each of the two groups;
* Compare patient satisfaction with meals in the two groups.

ELIGIBILITY:
Inclusion Criteria:

* Patient 65 years of age or older
* Patient not having objected to his participation in the study
* Patient affiliated to a social security scheme
* French-speaking patient

Exclusion Criteria:

* Patient receiving a diet with double portions (a side dish of vegetables and a side of starches)
* Patient receiving a diet not including a main course at dinner
* Patient receiving cold meals
* Patient receiving a controlled residue or fiber diet
* Patient receiving a diet with a modified texture: chopped, milled, mixed, semi-liquid or liquid
* Patient for whom weight cannot be measured
* Patient receiving partial or exclusive artificial nutrition (enteral or parenteral)
* Patient with a foreseeable length of stay of less than 6 days
* Patient with cognitive impairment
* Patient in accommodation in the care unit (risk of rapid transfer to the original department)
* For the second phase: patient who participated in the first phase of the study

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Each patient admitted to the internal medicine department will be included in the study, if he/she meets the inclusion criteria and does not present a excusion criterion.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2022-09-30 (Estimated); Primary Completion 2023-02-15 (Estimated); Study Completion 2023-02-15 (Estimated)

PRIMARY OUTCOMES:
Assessment of food intake | 6 days
  Evaluation of food intake between the two groups on day 6 ± 1 using the SEFI® tool: scale from 0 ("I don't eat anything at all") to 10 ("I eat normally") or visual evaluation portions consumed

CONTACTS AND LOCATIONS:
Overall Officials: Myriam SCELLES, Mrs, Principal Investigator — University Hospital, Caen

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Navarro DA, Boaz M, Krause I, Elis A, Chernov K, Giabra M, Levy M, Giboreau A, Kosak S, Mouhieddine M, Singer P. Improved meal presentation increases food intake and decreases readmission rate in hospitalized patients. Clin Nutr. 2016 Oct;35(5):1153-8. doi: 10.1016/j.clnu.2015.09.012. Epub 2015 Oct 9. PMID 26627844
- [Background] Hansen KV, Froiland CT, Testad I. Porcelain for All - a nursing home study. Int J Health Care Qual Assur. 2018 Aug 13;31(7):662-675. doi: 10.1108/IJHCQA-10-2016-0160. PMID 30354892
- [Background] Hiesmayr M, Schindler K, Pernicka E, Schuh C, Schoeniger-Hekele A, Bauer P, Laviano A, Lovell AD, Mouhieddine M, Schuetz T, Schneider SM, Singer P, Pichard C, Howard P, Jonkers C, Grecu I, Ljungqvist O; NutritionDay Audit Team. Decreased food intake is a risk factor for mortality in hospitalised patients: the NutritionDay survey 2006. Clin Nutr. 2009 Oct;28(5):484-91. doi: 10.1016/j.clnu.2009.05.013. Epub 2009 Jul 1. PMID 19573957
- [Background] Thibault R, Goujon N, Le Gallic E, Clairand R, Sebille V, Vibert J, Schneider SM, Darmaun D. Use of 10-point analogue scales to estimate dietary intake: a prospective study in patients nutritionally at-risk. Clin Nutr. 2009 Apr;28(2):134-40. doi: 10.1016/j.clnu.2009.01.003. Epub 2009 Feb 14. PMID 19223093